CLINICAL TRIAL: NCT06969001
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Administration of SCAI-005 Ophthalmic Solution in Healthy Korean Subjects
Brief Title: Clinical Study for the Evaluation of Safety and Tolerability of SCAI-005 Eye Drops
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCAI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: SCAI-005-101
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Wet Age Related Macular Degeneration
Keywords: axitinib; eyedrop; tyrosine kinase inhibitor; wetAMD; CNV; Phase1; SCAI-005

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental): Day 1: One time administration, 8 subjects randomized 3:1 to SCAI-005 or placebo in each cohort
  Interventions: Drug: SCAI-005 0.04% or placebo; Drug: SCAI-005 0.08% or placebo; Drug: SCAI-005 0.08% or placebo 2drops
- Multiple Ascending Dose (Experimental): Three times administration daily (TID) for 7days, 8 subjects randomized 3:1 to SCAI-005 or placebo in each cohort
  Interventions: Drug: SCAI-005 0.04% or placebo; Drug: SCAI-005 0.08% or placebo; Drug: SCAI-005 0.08% or placebo 2drops

INTERVENTIONS:
Drug: SCAI-005 0.04% or placebo — axitinib 0.014mg or placebo
Drug: SCAI-005 0.08% or placebo — axitinib 0.028mg or placebo
Drug: SCAI-005 0.08% or placebo 2drops — axitinib 0.056mg or placebo

SUMMARY:
To assess the single-dose and multiple-dose pharmacokinetics (PK), safety and tolerability of SCAI-005 eyedrops(axitinib) in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged 19 to 50 years at the time of screening
* Male subjects with a body weight of 55.0 kg or more, Female subjects with a body weight of 50kg or more, and within ±20% of ideal body weight at the time of screening
* Subject who voluntarily agrees to participate in this study and has given a written informed consent, after fully understanding the detailed explanation of this study

Exclusion Criteria:

* Subjects with symptoms suggestive of an acute disease at the time of screening
* Subjects with clinically significant and active diseases related to cardiovascular system, gastrointestinal system, respiratory system, endocrine system, neuropsychiatric system, hematologic/oncologic system
* Subjects meeting any of the following criteria based on examination during screening:

  1. AST, ALT > 1.5 X ULN
  2. Total bilitubin > 1.5 X ULN
  3. eGFR (estimated Glomerular Filtration Rate) < 90 mL/min/1.73 m2
  4. serological test result = positive
* Subjects with systolic blood pressure of 90 mmHg or less, or 150 mmHg or more, or diastolic blood pressure of 50 mmHg or less, or 100 mmHg or more after sitting for at least 5 minutes during screening (Visit 1)
* Subjects meeting any of the following criteria based on ophthalmological examination during screening:

  1. Best corrected visual acuity < 0.6
  2. IOP > 21 mmHg
  3. difference in IOP between both eyes > 4mmHg
  4. subjects who are assessed ineligible due to abnormal findings in other ophthalmonlogical examinations
* History or suspicion of conditions affecting visual organs such as keratitis, iritis, uveitis, retinitis, dry eye syndrome, strabismus within 12months prior to screening visit
* Ophthalmologic surgery within 12 months prior to screening visit
* Subjects with acute or chronic eye diseases requiring topical eyedrops at the time of screening
* Experience of adverse effects from contact lens use, or contact lens use within one month prior to screening visit, or inability to abstain from contact lens use during the clinical trial
* Subjects with a history of drug abuse or a positive result on a urine drug test at screening
* Subjects with a history of hypersensitivity to the investigational drug, or to drugs in the same class as the active ingredients
* Subjects who have participated in another clinical trial and received an investigational drug within 6 months prior to the anticipated first dose
* Subjects who have taken drug metabolism inducers or inhibitors, such as barbiturates, within one month prior to the expected first dosing date
* Subjects who have donated whole blood within 2 months, or component blood within 20 days
* Subjects who have taken any prescription drugs or oriental medicine within 2 weeks of the expected first dosing date, or any over-the-counter drugs or vitamins within 1 week of the expected first dosing date
* Subjects unable to restrict grapefruit or grapefruit-containing food consumption from 7 days prior to the anticipated first dose through the duration of the clinical trial.
* Subjects who regularly consume caffeine (e.g., coffee or green tea more than 5 units/day) or are unable to abstain from caffeine-containing foods from 24 hours prior to hospitalization to discharge
* Subjects who have consumed alcohol regularly (more than 210g/week) or are unable to abstain from alcohol from 24 hours prior to hospitalization to discharge
* Subjects who have regularly smoked (including e-cigarettes, more than 10 cigarettes/day) or are unable to abstain from 24 hours prior to hospitalization to discharge
* Female participants who are pregnant, or are breastfeeding
* Subjects who, during the entire clinical trial period and for at least 90 days after the last dose of the investigational drug, cannot or do not agree to use medically acceptable double contraception methods, or who do not agree to refrain from donating sperm during this period
* Subjects deemed unsuitable for participation by the investigator for other reasons

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation: Incidence, type, and severity of Adverse Events (AE) | 15days

OTHER OUTCOMES:
Cmax | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Single dose - Evaluation of pharmacokinetic profile
Tmax | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Single dose - Evaluation of pharmacokinetic profile
t1/2 | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Single dose - Evaluation of pharmacokinetic profile
CL/F | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Single dose - Evaluation of pharmacokinetic profile
AUClast | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Single dose - Evaluation of pharmacokinetic profile
Vz/F | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Single dose - Evaluation of pharmacokinetic profile
Cmax | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
Cmax,ss | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
Cmin,ss | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
Tmax | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
t1/2,ss | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
Tmax,ss | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
AUCtau,ss | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
Vz,ss/F | Pre-dose [day1, day3, day5, day8], 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile
CLss/F | Pre-dose, 10, 20, 30, 45 minutes, 1, 2, 4, 8, 12 hours after last administration
  Multiple dose - Evaluation of pharmacokinetic profile

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University, Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No